CLINICAL TRIAL: NCT06443398
Title: Evaluation of the Spine of Primary Caregivers of Children with Cerebral Palsy
Brief Title: Spine of Caregivers of Children with Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Dr. Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-T.ATAHAN-005
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy; Spine Deformity
Keywords: Primary Caregivers; Pain; Disability
MeSH Terms: conditions — Cerebral Palsy; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Primary caregivers with healthy children between the ages of 0-18 were included.
  Interventions: Other: There is no intervention in the study
- Study Group: Primary caregivers who had a child diagnosed with Cerebral Palsy between the ages of 0-18 and met the inclusion criteria were included.
  Interventions: Other: There is no intervention in the study

INTERVENTIONS:
Other: There is no intervention in the study — There is no intervention in the study

SUMMARY:
The purpose of this study was to assess pain (rest, activity, and night pain using the Visual Analog Scale), disability (neck using the Neck Disability Index; lumbar using the Oswestry Disability Index), and curvature (cervical, thoracic, and lumbar using the Spinal Mouse) in primary caregivers of children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver between the ages of 25-54
* Has a child diagnosed with Cerebral Palsy between the ages of 0-18
* Does not have inflammatory pain
* Without pain originating from abdominal-pelvic organs
* Volunteer caregivers were included

Exclusion Criteria:

* Having acute fracture and malignancy
* Had a surgical operation (related to spine disorders)
* Having a care burden for more than one disabled individual
* Caregivers with chronic illnesses (such as neurological, psychological disorders) were excluded

Ages: 25 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: It was conducted with caregivers of children with Cerebral Palsy who were receiving physiotherapy at Kırşehir Training and Research Hospital Physical Therapy and Rehabilitation Center and who met the exclusion-inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Life Quality | 16 week
  Parents' quality of life was measured using the Nottingham Health Profile. The scale has two parts. 0 represents the best health status, 100 the worst. Score on the scale and health status have an inverse relationship. As the score increases, the health status deteriorates.
Disability | 16 week
  Functional problems related to the neck were assessed using the Neck Disability Index. The scale has 10 items. There are 6 options in each item and each option is scored between 0 and 5 depending on the severity of the limitation. Although the total score of the survey varies between 0 and 50, a higher score indicates an increase in limitation.
Disability | 16 week
  Oswestry Disability Index was used to determine the degree of disability. The scale consists of a total of 10 items measuring the severity of pain, personal care, lifting, walking, sitting, standing, social life, sleeping, travel and pain degree. Each item is rated between 0-5. As the total score increases, the disability level increases. The maximum score is 50 points; Between 31 and 50 points is considered severe, between 11 and 30 points is considered moderate, and between 1 and 10 points is considered mild.
Spine | 16 week
  Spine evaluation was performed with a spinal mouse device. The device is a computer-aided electromagnetic device that can be held by hand and used to measure spinal mobility in various postures.

SECONDARY OUTCOMES:
Socio-demographic Form | 16 week
  Sociodemographic information of the caregivers, such as name, surname, age, gender, height, weight, BMI, and educational status, were recorded.
Pain Intensity | 16 week
  The pain intensity of the patients was measured using the Visual Analogue Scale. The pain intensity score ranges from 0 to 10. An increase in the score indicates an increase in pain; a decrease in the score indicates a decrease in pain.
Gross Motor Function Classification | 16 week
  Gross Motor Function Classification System (Children with Cerebral Palsy are classified in 5 levels (1-5) according to their motor skills, functional abilities, assistive technology and wheelchair requirements)

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No